CLINICAL TRIAL: NCT00680836
Title: Diarrhea-Predominant Irritable Bowel Syndrome in Persian Gulf Veterans
Brief Title: Gulf War Digestive Health Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GWRA-014-05F
Record Dates: First submitted 2008-05-16; First posted 2008-05-20 (Estimated); Results first posted 2014-08-29 (Estimated); Last update posted 2014-08-29 (Estimated); Status verified 2014-08

CONDITIONS: Irritable Bowel Syndrome; Small Intestinal Bacterial Overgrowth
Keywords: Irritable Bowel Syndrome; Diarrhea; Gulf War; Veterans; Small intestinal bacterial overgrowth (SIBO)
MeSH Terms: conditions — Irritable Bowel Syndrome; Diarrhea | interventions — Rifaximin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment Group (Active Comparator): These patients have IBS and are receiving the rifaximin.
  Interventions: Drug: Rifaximin
- Placebo group (Placebo Comparator): These patients have IBS and are receiving the placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — orally two times per day for 14 days
  Other Names: Inactive pill
  Arms: Placebo group
Drug: Rifaximin — 550 mg orally two times per day for 14 days
  Other Names: Xifaxan
  Arms: Treatment Group

SUMMARY:
The purposes of this study are to estimate the burden of disease due to chronic gastrointestinal illness in PG veterans, to evaluate whether Small Bowel Bacterial Overgrowth (SBBO) is associated with chronic diarrhea in PG veterans, and to determine whether eradication of SBBO reduces symptoms of chronic diarrhea, abdominal pain and bloating in PG veterans.

DETAILED DESCRIPTION:
Approximately 700,000 United States military personnel were deployed in the first Persian Gulf (PG) War. Several months after their return, up to 25% of Veterans had persistent symptoms which they suspected were related to their military service in the Gulf. Among the most frequent were gastrointestinal symptoms such as loose stools, excessive gas and abdominal pain. These symptoms are typical of diarrhea-predominant irritable bowel syndrome (IBS).

The cause of IBS is not known; speculated mechanisms include altered GI motility, bacterial overgrowth, visceral hypersensitivity and psychological stress. Another proposed mechanism relates to the fact that up to one third of patients with IBS describe the onset of their symptoms following acute gastroenteritis. This is called post-infective IBS (PI-IBS). How acute gastroenteritis leads to persistent GI symptoms of IBS is not known. A limited amount of data suggests that patients with IBS may have an imbalance in their gastrointestinal microflora. Several studies indicate that small bowel bacterial overgrowth is more common in individuals with IBS. Symptoms of SBBO are similar to diarrhea-predominant IBS and include chronic diarrhea, bloating and abdominal pain.

More than 50 percent of military personnel developed acute gastroenteritis while on duty in the Gulf. Most of them who reported symptoms of IBS had an acute onset which occurred in association with an episode of acute gastroenteritis during their tour of duty. Other travelers are known to be colonized by new micro-organisms during travel to foreign countries. This acquisition is thought to be related to a change in diet. The natural history of this change in bowel flora, in part, depends on host factors and can persist for months after travel abroad. It seems likely, that PG veterans with persistent diarrhea and a negative work-up for known GI diseases have PI-IBS. No study in the past has evaluated the role of SBBO in causing chronic GI symptoms in PG Veterans. Furthermore, soldiers involved in combat are exposed to a highly stressful environment, perhaps making them more susceptible to persistent symptoms.

We hypothesize that PG veterans with chronic GI symptoms have symptoms of diarrhea predominant IBS and this is caused by SBBO due to a change in microflora during deployment in the Persian Gulf and that it is predisposed to by the stress of combat. Intestinal microflora, once altered, is known to be relatively stable; once mucosal damage occurs it may become permanent.

Objectives Objective # 1: Estimate the burden of disease due to chronic gastrointestinal illness in PG veterans.

Hypothesis:

i. The prevalence of GI symptoms is high in PG veterans. ii. The prevalence of IBS is higher in veterans who report acute gastroenteritis during the period of deployment.

iii. PG Veterans with IBS have a lower IBS related QOL

Objective # 2: Evaluate whether SBBO is associated with chronic diarrhea in PG veterans.

Hypothesis i. SBBO is more common in PG veterans than non deployed veterans. ii. SBBO is more common in PG veterans with diarrhea-predominant IBS vs. those without.

Objective: # 3: Determine whether eradication of SBBO reduces symptoms of chronic diarrhea, abdominal pain and bloating in PG Veterans.

Hypothesis:

i. Treatment with rifaximin, a non-absorbable antibiotic, will improve symptoms and QOL in Veterans with SBBO.

ELIGIBILITY:
Inclusion Criteria:

* Men and women age 32-75 years
* Rome III criteria for diarrhea-predominant IBS
* Symptom onset after an apparent episode of acute gastroenteritis
* Symptoms of > 3 months duration
* Normal endoscopic appearance of the colonic mucosa
* Negative markers for celiac disease and inflammatory bowel disease.
* Normal thyroid function and serum calcium levels.
* Must have served in the military or reserves during the time of Operation Desert Storm (August 1990 to May 1991)

Exclusion Criteria:

* Clinically significant cardiac, pulmonary, hepatic or renal dysfunction
* History of/or presence of systemic malignancy
* Current evidence of any gastrointestinal disorder such as celiac disease or inflammatory bowel disease (i.e. Crohns disease or ulcerative colitis)
* Current effects of drug or alcohol abuse
* Investigator perception of patients inability to comply with study protocol
* Unstable psychiatric disease
* Recent change in gastrointestinal medications
* Subjects with a positive pregnancy test
* Subject is currently participating in another research protocol that could interfere or influence the outcome measures of the present study

Ages: 35 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2007-10; Primary Completion 2008-10 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ashok K Tuteja, MD MPH, Principal Investigator — Division of Epidemiology
Locations (1):
- Division of Epidemiology, Salt Lake City, Utah, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo Group: These patients have Irritable Bowel syndrome and are receiving the placebo twice a day
- Active Group: These patients have Irritable Bowel syndrome and are receiving rifaximin 550mg twice a day
Period: Overall Study
Arm/Group | Placebo Group | Active Group
Started | 27 | 27
Completed | 19 | 25
Not Completed | 8 | 2
Not completed — Withdrawal by Subject | 3 | 0
Not completed — Lost to Follow-up | 3 | 1
Not completed — Physician Decision | 2 | 1

BASELINE CHARACTERISTICS:
Population: A total of 54 patients were randomized. Of that 54 patients,10 patients were excluded from the analyses. Reasons included, patient withdrawal, physician decision, and loss to follow up.Total of 44 patients were analysed. All data presented here, includes the 44 patients only.
Groups:
- Placebo: These patients have Irritable Bowel syndrome (IBS) and are receiving the placebo twice a day
- Treatment: These patients have Irritable Bowel syndrome (IBS) and are receiving the rifaximin 550mg twice a day
- Total: Total of all reporting groups
Arm/Group | Placebo | Treatment | Total
Number analyzed (Participants) | 19 | 25 | 44
Age, Customized [Mean (Full Range); unit: years] | 52 [41 to 67] | 56 [33 to 77] | 52 [33 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 5 | 6
  Male | 18 | 20 | 38
Region of Enrollment [Number; unit: participants]
  United States | 19 | 25 | 44

OUTCOME MEASURES:

1. Primary Outcome: Global Improvement Scale
Description: Improvement in Irritable Bowel Syndrome symptoms post treatment is measured. This scale is not measured at baseline. Participants are asked if their symptoms improved or got worse and to rate it on a scale of 1- 7 for seven days. Average score for 7 days is calculated. The Global improvement scale ranges from 1- 7. Score of 1-3 means the IBS symptoms got worse, 4 means no change and 5-7 means improvement in the IBS symptoms.
Time Frame: Measured for seven days at the end of 2 weeks treatment and average score is calculated
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Placebo Group: These patients have IBS and are receiving placebo tablets twice a day
- Active Group: These patients have IBS and are receiving the rifaximin 550mg twice a day
Arm/Group | Placebo Group | Active Group
Number analyzed (Participants) | 19 | 25
units on a scale | 4.3 (1.0) | 4.3 (0.9)
Statistical Analysis 1: Comparison: Placebo Group vs Active Group; Test type: Superiority or Other; p = 0.26, t-test, 2 sided; Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-1.0 to 0.3]

2. Secondary Outcome: Change in Stool Frequency (Number of Bowel Movements Per Day)
Description: Change in stool frequency (number of bowel movements per day) compared from baseline to post treatment is measured. Number of bowel movements per day before treatment is subtracted from the number of bowel movements per day after treatment. The change in frequency has been reported in the outcomes table.
Time Frame: 2 weeks
Measure: Mean (95% Confidence Interval); unit: Bowel movements/ day
Groups:
- Placebo Group: These patients have IBS and are receiving the placebo twice a day
Arm/Group | Placebo Group | Active Group
Number analyzed (Participants) | 19 | 25
Bowel movements/ day | -0.3 [-0.7 to 0.2] | -0.1 (0.2) [-0.4 to 0.2]
Statistical Analysis 1: Comparison: Placebo Group vs Active Group; Test type: Superiority or Other; p = 0.98, t-test, 2 sided; Mean Difference (Final Values) = 0.0, 95% CI 2-sided [0.0 to 0.5]

3. Secondary Outcome: Change in Stool Consistency
Description: Change in Stool consistency from baseline to post treatment is measured. Bristol stool scale is used for this purpose. The scale ranges from a value of 1- 7; 1 being very hard stool to 7 being liquid stools. The change is measured for 1 week post-treatment and the average consistency is used for the purpose of measuring change from baseline.
Time Frame: 2 weeks
Measure: Mean (95% Confidence Interval); unit: units on a scale (BSS)
Arm/Group | Placebo Group | Active Group
Number analyzed (Participants) | 19 | 25
units on a scale (BSS) | -0.4 (0.2) [-0.9 to 0.1] | -0.3 (0.2) [-0.7 to 0.1]
Statistical Analysis 1: Comparison: Placebo Group vs Active Group; Test type: Superiority or Other; p = 0.78, t-test, 2 sided; Mean Difference (Final Values) = 0.1

4. Secondary Outcome: Change in Bowel Urgency
Description: Urgency in a bowel movements compared from baseline to post treatment was measured. Participants were asked to note if they had urgency at bowel movements (meaning if they had to rush to the restroom). They marked either 'yes' or 'no'. The percentage of the time they said yes was calculated for 7 days. The difference between baseline and post treatment urgency was calculated.
Time Frame: 2 weeks
Measure: Mean (95% Confidence Interval); unit: difference in percentage of 'Yes'
Arm/Group | Placebo Group | Active Group
Number analyzed (Participants) | 19 | 25
difference in percentage of 'Yes' | 0.0 (0.1) [-0.2 to 0.2] | -0.1 (0.1) [-0.3 to 0.1]
Statistical Analysis 1: Comparison: Placebo Group vs Active Group; Test type: Superiority or Other; p = 0.64, Chi-squared; Mean Difference (Final Values) = 0.0, 95% CI 2-sided [-0.2 to 0.2]

5. Secondary Outcome: Change in Abdominal Pain With Bowel Movement
Description: Severity of abdominal pain on a scale of 0 to 4 was measured; 0 meaning no pain to 4 meaning severe pain. Change in abdominal pain from baseline to post treatment was calculated.
Time Frame: 2 weeks
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo Group | Active Group
Number analyzed (Participants) | 19 | 25
units on a scale | -0.3 (0.2) [-0.9 to 0.3] | -0.2 (0.2) [-0.6 to 0.2]
Statistical Analysis 1: Comparison: Placebo Group vs Active Group; Test type: Superiority or Other; p = 0.72, t-test, 2 sided; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-0.7 to 0.5]

6. Secondary Outcome: Change in Bloating
Description: Bloating is measured on a scale from 0 to 4; 0 = no bloating to 4 = severe bloating. Change in bloating is calculated from baseline to post treatment.
Time Frame: 2 weeks
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo Group | Active Group
Number analyzed (Participants) | 19 | 25
units on a scale | -0.2 (0.2) [-0.7 to 0.3] | -0.2 (0.2) [-0.7 to 0.3]
Statistical Analysis 1: Comparison: Placebo Group vs Active Group; Test type: Superiority or Other; p = 0.86, t-test, 2 sided; Mean Difference (Net) = 0.0, 95% CI 2-sided [-0.5 to 0.6]

ADVERSE EVENTS:
Time Frame: The participants were followed up for 6 months after treatment ended.
Arm/Group | Placebo Group | Active Group
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/27
Other Adverse Events (participants affected / at risk) | 10/27 | 14/27
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Group (N=27) | Active Group (N=27)
accidental Injury (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 3 (3)
Bloating (Gastrointestinal disorders) | 1 (1) | 2 (2)
Infection (Infections and infestations) | 1 (1) | 3 (3)
Anxiety (Nervous system disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Surgery (Surgical and medical procedures) | 1 (1) | 5 (5)
Body Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No